CLINICAL TRIAL: NCT06550193
Title: The Use of Augmented Reality (AR) or Virtual Reality (VR) to Enhance the Precision and Accuracy of Ultrasound-guided Medical Procedures
Brief Title: AR/VR for Ultrasound-guided Medical Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean-Louis Horn, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 75204
Record Dates: First submitted 2024-07-16; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Augmented Reality; Virtual Reality
Keywords: ultrasound-guided procedure; nerve block

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention, which involves utilizing AR/VR technology during ultrasound-guided procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AR/VR (Experimental): AR/VR technology for ultrasound-guided procedures.
  Interventions: Device: Ultrasound-guided procedure using AR/VR technology

INTERVENTIONS:
Device: Ultrasound-guided procedure using AR/VR technology — Participants will receive the intervention, which involves utilizing AR/VR technology during ultrasound-guided procedures (e.g., regional anesthesia, line placement). All participants will receive standard pre- and post-block or line care as they normally would for the ultrasound-guided procedure.

SUMMARY:
The study seeks to assess the efficacy of incorporating augmented reality (AR) or virtual reality (VR) technology into ultrasound-guided medical procedures such as regional anesthesia and line placement. By utilizing AR/VR devices, the investigators will improve the ergonomics when using ultrasound to guide procedures. The aims are to enhance visualization of anatomical structures and improve procedural accuracy for clinicians. The study aims to evaluate the feasibility, and effectiveness of integrating AR/VR technology into ultrasound-guided procedures, with the ultimate goal of improving patient outcomes.

DETAILED DESCRIPTION:
The investigators aim to learn several key insights from this study. Firstly, they hope to determine the extent to which augmented reality (AR) or virtual reality (VR) technology can enhance the precision and accuracy of ultrasound-guided medical procedures, such as regional anesthesia and line placement. This includes evaluating whether AR/VR visualization leads to improved needle placement and reduced complication rates.

Furthermore, the investigators aim to evaluate the usability and acceptance of AR/VR technology among clinicians, considering factors such as user experience, comfort, and integration with existing workflow processes.

The importance of this new knowledge lies in its potential to improve medical practice by leveraging cutting-edge technology to improve patient outcomes and expand access to quality healthcare globally. If AR/VR proves to be effective in enhancing procedural accuracy, it could lead to significant advancements in healthcare delivery, particularly in underserved communities and resource-limited settings by leveraging remote care. Additionally, insights gained from this study could inform the development of future AI assisted AR/VR applications in medicine, driving innovation and improving the standard of care across various medical specialties.

ELIGIBILITY:
Inclusion Criteria:

* adult patients presenting for ultrasound-guided procedures, with ASA physical status I, II, or III.

Exclusion Criteria:

* pregnancy
* incarceration
* BMI >35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Procedure success rate (Primary Block) | Document the block result pre-operatively (at least 30 min following block completion), or within one hour upon arriving to PACU
  Document the block result in pre-op, if feasible, or PACU by testing sensory (cold spray) and motor function on all nerves covered by the block
Post-operative opioid consumption | 12 hours after surgery
  Morphine milligram equivalents (MME) will be measured post-operatively
Post-operative pain scores | 12 hours after surgery
  Trend pain scores on 11-point NRS scale (from 0 to 10) following the procedure

SECONDARY OUTCOMES:
Clinician satisfaction | Within 24 hours of block completion
  A short survey will be utilized to gather data on clinicians' perceptions of the ease of use, effectiveness, and overall experience with AR/VR tools compared to traditional methods.
Procedure duration | During the procedure
  Time of procedure from initial needle insertion to needle removal will be calculated
Needle pass/redirection | During the procedure
  The number of times a clinician must remove the needle from the patient completely and reattempt will be calculated.
Needle visualisation | Within 24 hours of block completion
  A subjective score will be assessed on a short survey to clinicians.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No